CLINICAL TRIAL: NCT05912179
Title: Prospective Single Centre Observational Study to Compare the Diagnostic Yield of Different Modalities of Liver Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Suresh Vasan Venkatachalapathy, Consultant Hepatologist, Nottingham University Hospitals NHS Trust
Other Study IDs: 22-577C
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Liver Diseases; Liver Fibrosis
Keywords: EUS; Endoscopic Ultrasound; Liver Biopsy; Percutaneous liver biopsy; Trans-jugular liver biopsy; EUS shear wave measurement
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — liver biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EUS guided liver biopsy: Patients having liver biopsy through endoscopic ultrasound technique
  Interventions: Diagnostic Test: liver biopsy - EUS guided
- Percutaneous liver biposy: Patients having liver biopsy percutaneously
  Interventions: Diagnostic Test: Liver biopsy - percutaneous
- Transjugular liver biopsy: Patients having liver biopsy via a transjugular route
  Interventions: Diagnostic Test: Liver biopsy - transjugular

INTERVENTIONS:
Diagnostic Test: Liver biopsy - percutaneous — liver biopsy obtained using percutaneous ultrasound guided technique
  Groups: Percutaneous liver biposy
Diagnostic Test: Liver biopsy - transjugular — liver biopsy obtained using an interventional transjugular approach
  Groups: Transjugular liver biopsy
Diagnostic Test: liver biopsy - EUS guided — liver biopsy obtained during endoscopic ultrasound
  Groups: EUS guided liver biopsy

SUMMARY:
The goal of this study is to learn about endoscopic ultrasound(EUS) guided liver biopsy and how this compares to traditional methods of obtaining liver biopsy samples, in patients with liver disease.

The main questions it aims to answer are:

1. is EUS liver biopsy equally as good as other types of techniques
2. are there any advantages to using the EUS technique to obtain liver biopsies Researchers will compare data from patients who have had a liver biopsy with a traditional technique with those who have undergone EUS-guided biopsy.

DETAILED DESCRIPTION:
Introduction:

The rising incidence of liver disease (LD) has led to an increased demand on services for accurate and prompt diagnosis and staging, to facilitate treatments and early interventions. While non-invasive diagnostic tests (e.g. transient elastography, ELF biomarkers) are the standard of care to stratify fibrosis burden, there are still cases that require a liver biopsy (LB) for assessment of fibrosis and aetiology of disease. Traditional methods such as percutaneous LB (PLB) and transjugular LB (TJLB) are well established, however there is a recognised burden on the services, translating to prolonged waiting times and delays in diagnosis. Endoscopic ultrasound-guided liver biopsy (EUS-LB) is emerging as a novel, minimally invasive way of not only securing a tissue sample, but also providing an in-depth assessment of other parameters such as portal pressure gradient (PPG), shearwave measurement (SWM) and varices assessment. The aim of this study was to test the diagnostic adequacy, fibrosis staging, length of stay post procedure and complication rates following the above modalities of Liver biopsy.

Methods:

This is a single centre prospective observational study to assess the diagnostic accuracy of liver biopsy through different modalities. Data will be as collected prospectively from all adult patients patients undergoing any form of LB in a single tertiary hospital for 12 months:September 2022 to September 2023. Information was collected will be on demographics, biopsy indication, length of core, length of stay (LoS), complications and diagnostic yield.

Primary aim: To assess the diagnostic yield of liver biopsy through EUS-LB, Trans-jugular liver biopsy and percutaneous ultrasound guided liver biopsy.

Secondary aim;

1. Technical success rate,
2. Length of the cores obtained
3. Number of portal tracts
4. Accuracy of Shear wave measurement compared to Liver biopsy
5. complications rate
6. Length of stay

Dissemination plan:

the results of the study will be disseminated through presentation at national/ international meetings and publishing in peer reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* underwent liver biopsy either through EUS, percutaneous or transjugular route

Exclusion Criteria:

- under 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective observation of all consecutive adult patients undergoing Liver biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with adquate tissue to make accurate diagnosis with different modalities of Liver biopsy | 1 year
  patient in whom a diagnosis has been reached or supported by histological results

SECONDARY OUTCOMES:
Length of stay | 1 year
  length of stay of patients undergoing different Liver biopsy modalities
Complication rate with different modalities | 30 days
  complication rate of different modalities of liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Vasan Suresh Vasan, Principal Investigator — Nottingham University Hospitals
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD